CLINICAL TRIAL: NCT02612168
Title: Effectiveness of an Image Analysing Algorithm to Diagnose Melanoma Compared to Gold Standard Histological Determination
Brief Title: Melanoma Image Analysis Algorithm (MIAA) Validation Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Skin Analytics Limited (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: SA-001-4ev
Record Dates: First submitted 2015-11-18; First posted 2015-11-23 (Estimated); Last update posted 2019-01-25 (Actual); Status verified 2019-01

CONDITIONS: Malignant Melanoma
Keywords: Diagnosis; skin imaging
MeSH Terms: conditions — Melanoma; Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- All patients (Experimental): Each patient will have any pigmented lesions (PLs) which are due to be biopsied, two PLs not due for biopsy and one patch of healthy skin photographed. Each will be photographed using three cameras: A standard DSLR and two smartphones with a dermoscopic lens attachment. Photographic images will be analysed by Melanoma Image Analysis Algorithm (MIAA)
  Interventions: Device: Melanoma Image Analysis Algorithm (MIAA)

INTERVENTIONS:
Device: Melanoma Image Analysis Algorithm (MIAA) — The images will be analysed by MIAA (Melanoma Image Analysis Algorithm). The MIAA result for PLs that are biopsied will be compared to the diagnosis made from the biopsy. The MIAA result for PLs not biopsied will be compared to clinician diagnosis.

SUMMARY:
Prospective, single-arm, cross-sectional, study to establish the effectiveness of MIAA to detect melanoma in pigmented lesions, compared to gold standard histological determination.

DETAILED DESCRIPTION:
Skin Analytics Limited have developed an algorithm (MIAA) which reviews photographs of pigmented lesions to determine whether melanoma is likely to be present. This study aims to establish how well MIAA determines the presence or absence of melanoma, compared to a biopsy.

Pigmented lesions that a dermatologist has decided to biopsy, and are suitable for photographing, will be photographed up to five times in a single visit. Three different camera will be used, and two different dermoscopic lens attachments will be used on smartphone cameras. Images will be analysed by MIAA and the results compared to the biopsy result. Clinicians, patients and the statistical analysis team will be blinded to the result of MIAA.

At least 65 pigmented lesions positive for melanoma (as determined by biopsy) are required, which is predicted to mean 1250 patients will be recruited.

ELIGIBILITY:
Inclusion Criteria:

* Participant is willing and able to give informed consent for participation in the study,
* Male or Female, aged 18 years or above,
* Have at least 1 lesion suitable for photographing that is scheduled for biopsy to determine the presence of melanoma,
* In the Investigators opinion, able and willing to comply with all study requirements.

Exclusion Criteria:

• Any other significant disease or disorder which, in the opinion of the Investigator, may either put the participants at risk because of participation in the study, or may influence the result of the study, or the participant's ability to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 514 (Actual)
Dates: Start 2017-01-11 (Actual); Primary Completion 2018-07-11 (Actual); Study Completion 2018-07-11 (Actual)

PRIMARY OUTCOMES:
The Area Under the Curve of a Receiver Operating Characteristic (AUROC) curve of MIAA result, using a maximum likelihood estimation (MLE) from all of the available images of biopsied lesions, compared to the biopsy result | Study completion, on average 2 weeks
  Compare the MIAA result with the biopsy result

SECONDARY OUTCOMES:
The sensitivity of MIAA, using a MLE from all of the available images of biopsied lesions, compared to the biopsy result | Study completion, on average 2 weeks
  %true positives, as determined by biopsy, identified
The sensitivity of MIAA, using a MLE from all of the available images of non-biopsied lesions, compared to clinical assessment | Study completion, on average 2 weeks
  %true positives, as determined by clinician, identified
The specificity of MIAA, using a MLE from all of the available images of biopsied lesions, compared to the biopsy result | Study completion, on average 2 weeks
  %true negatives, as determined by biopsy, identified
The specificity of MIAA, using a MLE from all of the available images of non-biopsied lesions, compared to clinical assessment | Study completion, on average 2 weeks
  %true negatives, as determined by clinician, identified
The positive predictive value of MIAA, using a MLE from all of the available images of biopsied lesions, compared to the biopsy result | Study completion, on average 2 weeks
  Probability that subjects with a positive MIAA result have a positive biopsy result
The positive predictive value of MIAA, using a MLE from all of the available images of non-biopsied lesions, compared to clinical assessment | Study completion, on average 2 weeks
  Probability that subjects with a positive MIAA result are thought likely to have melanoma by the clinician
The negative predictive value of MIAA, using a MLE from all of the available images of biopsied lesions, compared to the biopsy result | Study completion, on average 2 weeks
  Probability that subjects with a negative MIAA result have a negative biopsy result
The negative predictive value of MIAA, using a MLE from all of the available images of non-biopsied lesions, compared to clinical assessment | Study completion, on average 2 weeks
  Probability that subjects with a negative MIAA result are not thought likely to have melanoma by the clinician
The false positive rate of MIAA, using a MLE from all of the available images of biopsied lesions, compared to the biopsy result | Study completion, on average 2 weeks
  Probability that subject with positive MIAA result has a negative biopsy result
The false positive rate of MIAA, using a MLE from all of the available images of non-biopsied lesions, compared to clinical assesment | Study completion, on average 2 weeks
  Probability that subject with positive MIAA result are not thought likely to have melanoma by the clinician
The false negative rate of MIAA, using a MLE from all of the available images of biopsied lesions, compared to the biopsy result | Study completion, on average 2 weeks
  Probability that subject with negative MIAA result has a positive biopsy result
The false negative rate of MIAA, using a MLE from all of the available images of non-biopsied lesions, compared to clinical assessment | Study completion, on average 2 weeks
  Probability that subject with negative MIAA result are thought likely to have melanoma by the clinician
The AUROC of MIAA, using images of biopsied lesions from each of the image capture apparatus combinations, compared to the biopsy result | Study completion, on average 2 weeks
  Comparing the MIAA result, using images taken by each device, with the biopsy result
The AUROC of MIAA, using images of non-biopsied lesions from each of the image capture apparatus combinations, compared to clinical assessment | Study completion, on average 2 weeks
  Comparing the MIAA result, using images taken by each device, with the clinician's diagnosis
The sensitivity of MIAA, using images of biopsied lesions from each of the image capture apparatus, compared to the biopsy result | Study completion, on average 2 weeks
  %true positives, as determined by biopsy, identified by each imaging device
The sensitivity of MIAA, using images of non-biopsied lesions from each of the image capture apparatus, compared to clinical assessment | Study completion, on average 2 weeks
  %true positives, as determined by clinician, identified by each imaging device
The specificity of MIAA, using images of biopsied lesions from each of the image capture apparatus, compared to the biopsy result | Study completion, on average 2 weeks
  %true negatives, as determined by biopsy, identified by each imaging device
The specificity of MIAA, using images of non-biopsied lesions from each of the image capture apparatus, compared to clinical assessment | Study completion, on average 2 weeks
  %true negatives, as determined by clinician, identified by each imaging device
The positive predictive value of MIAA, using images of biopsied lesions from each of the image capture apparatus, compared to the biopsy result | Study completion, on average 2 weeks
  Probability that subjects with a positive MIAA result, using images taken by each device, have a positive biopsy result
The positive predictive value of MIAA, using images of non-biopsied lesions from each of the image capture apparatus, compared to clinical assessment | Study completion, on average 2 weeks
  Probability that subjects with a positive MIAA result, using images taken by each device, are thought likely to have melanoma by the clinician
The negative predictive value of MIAA, using images of biopsied lesions from each of the image capture apparatus, compared to the biopsy result | Study completion, on average 2 weeks
  Probability that subjects with a negative MIAA result, using images taken by each device, have a negative biopsy result
The negative predictive value of MIAA, using images of non-biopsied lesions from each of the image capture apparatus, compared to clinical assessment | Study completion, on average 2 weeks
  Probability that subjects with a negative MIAA result, using images taken by each device, are not thought likely to have melanoma by the clinician
The false positive rate of MIAA, using images of biopsied lesions from each of the image capture apparatus, compared to the biopsy result | Study completion, on average 2 weeks
  Probability that subject with positive MIAA result, using images taken by each device, has a negative biopsy result
The false positive rate of MIAA, using images of non-biopsied lesions from each of the image capture apparatus, compared to clinical assessment | Study completion, on average 2 weeks
  Probability that subject with positive MIAA result, using images taken by each device, are not thought likely to have melanoma by the clinician
The false negative rate of MIAA, using images of biopsied lesions from each of the image capture apparatus, compared to the biopsy result | Study completion, on average 2 weeks
  Probability that subject with negative MIAA result, using images taken by each device, has a positive biopsy result
The false negative rate of MIAA, using images of non-biopsied lesions from each of the image capture apparatus, compared to clinical assessment | Study completion, on average 2 weeks
  Probability that subject with negative MIAA result, using images taken by each device, are thought likely to have melanoma by the clinician
The concordance of MIAA result between each of the image capture apparatus | Study completion, on average 2 weeks
  The extent to which the image capture apparatus generate the same MIAA results as the other devices
The number of adverse events, including adverse device events and serious adverse events. | Study completion, on average 2 weeks
  The number of adverse events, including adverse device events and serious adverse events.
The proportion of lesions with 4 images that can be analysed by MIAA | Study completion, on average 2 weeks
  The proportion of lesions with 4 images that can be analysed by MIAA
The proportion of lesions with at least 1 readable images that can be analysed by MIAA, | Study completion, on average 2 weeks
  The proportion of lesions with at least 1 readable images that can be analysed by MIAA,
The AUROC curve of the MIAA result, using MLE from all of the available images of non-biopsied PLs, compared to the clinical assessment | Study completion, on average 2 weeks
  Compare the MIAA result with the clinicians assessment

OTHER OUTCOMES:
Impact of patient characteristics on the AUROC assessment of MIAA | Study completion, on average 2 weeks
  A statistical model will test the whether patient characteristics, such as age, gender, and skin type, affect the overall result and if so by how much
Impact of the image variables on the AUROC assessment of MIAA | Study completion, on average 2 weeks
  A statistical model will test the whether image variables, such as manufacturer and lens type, affect the overall result and if so by how much
Impact of the assessing clinician's level of experience on the AUROC assessment of MIAA | Study completion, on average 2 weeks
  A statistical model will test the whether the clinicians' level of experience affect the overall result and if so by how much
The concordance between the referring clinician's level of confidence for biopsy and the MIAA result | Study completion, on average 2 weeks
  The extent to which the clinician's assessment of melanoma is the same as biopsy and MIAA results

CONTACTS AND LOCATIONS:
Overall Officials: Ioulios Palamaras, MD PhD, Principal Investigator — Royal Free London NHS Foundation Trust
Locations (7):
- United Kingdom (7):
  - Royal Devon and Exeter, Exeter, Devon
  - Whipps Corss Hospital, Leytonstone, London
  - Royal Stoke University Hospital, Stoke, Staffordshire
  - Russells Hall Hospital, Dudley, West Midlands
  - Bristol Royal Infirmary, Bristol
  - Royal Free London NHS Foundation Trust, London
  - Churchill Hospital, Oxford

IPD SHARING:
Plan to Share IPD: Undecided